CLINICAL TRIAL: NCT00679419
Title: Coronary Artery Disease and Renal Failure Registry
Acronym: CAD-REF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut für Klinisch-Kardiovaskuläre Forschung GmbH (Network)
Collaborators: BMBf (Federal Ministry of Education and Research) (Unknown); KfH Kuratorium für Dialyse und Nierentransplantation e.V. (Unknown); Amgen (Industry); AstraZeneca (Industry); Boehringer Ingelheim (Industry); Sanofi (Industry)
Other Study IDs: 1-071812
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease; Renal Failure
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Urine, whole blood, serum

GROUPS / COHORTS (6):
- Group 0 (Controllgroup): eGFR >= 90 ml/min/1.73m^2 and no proteinuria
- Group 1: eGFR >= 90 ml/min/1.73m^2 and proteinuria
- Group 2: eGFR 60 - 89 ml/min/1.73m^2
- Group 3: eGFR 30 - 59 ml/min/1.73m^2
- Group 4: eGFR 15 - 29 ml/min/1.73m^2
- Group 5: eGFR < 15 ml/min/1.73m^2 or requiring dialysis

SUMMARY:
It is the aim of the multi-centric and prospective registry to analyze in patients with CAD the impact of different grades of renal failure on the outcome and course of the patients and to correlate these with clinical variables.

In particular, the registry has the following objectives:

* prospective consecutive assessment of all patients with coronary artery disease and renal failure in the participating hospitals of the registry
* evaluation of the outcome and course of patients with regard to their different stages of renal failure at baseline
* analysis of the impact of different therapeutic strategies on acute and long-term outcomes
* identification of clinical risk factors, novel biomarkers and genetic markers for an unfavorable long-term outcome

ELIGIBILITY:
Inclusion Criteria:

* Women and men >= 18 years of age
* Patients with actually performed interventional coronary angiography and there a documented coronary heart disease, defined as at least one documented stenosis >= 50 % in at least one main coronary vessel (Main steam; RCX; RIVA; RCA)
* European/Caucasian descent (European/Caucasian parents and grandparents)
* Availability of an urine, serum- and EDTA blood sample of the patient
* Documented consent of patients for handling of personal medical data, including a genetic analysis

Exclusion Criteria:

* Patients who have been already recruited into this registry
* Patients with organ transplantations, apart from kidney transplantations
* Immunosuppressive therapy, apart from immunosuppressive therapy after kidney transplantation
* Patients with polycystic renal disease
* Pregnant and breastfeeding patients
* Known malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed coronary artery disease were consecutively enrolled and classified into six groups according to their kidney function
Sampling Method: Non-Probability Sample
Enrollment: 3352 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-05 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | two years

SECONDARY OUTCOMES:
manner of death | two years
  cardiac death; non-cardiac death; death of unknown cause

OTHER OUTCOMES:
Interventions | two years
  Myocardial infarction or stroke; Renal failure or contrast medium induced nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Eva Brand, Prof. Dr., Principal Investigator — University Hospital of Muenster; Holger Reinecke, Prof. Dr., Principal Investigator — University Hospital of Muenster; Günter Breithardt, Prof. Dr., Principal Investigator — University Hospital of Muenster; Hermann Pavenstädt, Prof. Dr., Principal Investigator — University Hospital of Muenster
Locations (32):
- Germany (32):
  - Universitätsklinikum Aachen, Aachen
  - Zentralklinik Bad Berka, Bad Berka
  - Herz- und Gefäßklinik Bad Neustadt, Bad Neustadt an der Saale
  - Schüchtermann-Klinik, Bad Rothenfelde
  - Herzzentrum Brandenburg, Brandenburg
  - St.-Vincenz-Hospital, Coesfeld
  - Klinikum Lippe-Detmold, Detmold
  - Herzzentrum Duisburg, Duisburg
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Alfried Krupp Krankenhaus Essen, Essen
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Universitätsklinikum Halle/Saale, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - St. Marienhospital Hamm, Hamm
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Privatklinik Dr. Schindlbeck, Herrsching am Ammersee
  - Herzzentrum Lahr, Lahr
  - Kardiologische Praxis Dr. Schön, Mühldorf
  - Klinik Augustium München, München
  - Klinikum Neuperlach, München
  - Raphaelsklinik Münster, Münster
  - St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster, Münster
  - Lukaskrankenhaus Neuss, Neuss
  - Euregioclinic Nordhorn, Nordhorn
  - St. Vincenz-Krankenhaus, Paderborn
  - Klinikum Pirna, Pirna
  - Christliches Krankenhaus Quakenbrück e.V., Quakenbrück
  - Zentralklinikum Suhl, Suhl
  - Josephs-Hospital Warendorf, Warendorf

REFERENCES:
- [Derived] Engelbertz C, Pinnschmidt HO, Freisinger E, Reinecke H, Schmitz B, Fobker M, Schmieder RE, Wegscheider K, Breithardt G, Pavenstadt H, Brand E. Sex-specific differences and long-term outcome of patients with coronary artery disease and chronic kidney disease: the Coronary Artery Disease and Renal Failure (CAD-REF) Registry. Clin Res Cardiol. 2021 Oct;110(10):1625-1636. doi: 10.1007/s00392-021-01864-5. Epub 2021 May 26. PMID 34036426
- [Derived] Engelbertz C, Reinecke H, Breithardt G, Schmieder RE, Fobker M, Fischer D, Schmitz B, Pinnschmidt HO, Wegscheider K, Pavenstadt H, Brand E. Two-year outcome and risk factors for mortality in patients with coronary artery disease and renal failure: The prospective, observational CAD-REF Registry. Int J Cardiol. 2017 Sep 15;243:65-72. doi: 10.1016/j.ijcard.2017.05.022. Epub 2017 May 7. PMID 28526542
- [Derived] Brand E, Pavenstadt H, Schmieder RE, Engelbertz C, Fobker M, Pinnschmidt HO, Wegscheider K, Breithardt G, Reinecke H. The Coronary Artery Disease and Renal Failure (CAD-REF) registry: trial design, methods, and aims. Am Heart J. 2013 Sep;166(3):449-56. doi: 10.1016/j.ahj.2013.06.010. Epub 2013 Jul 23. PMID 24016493
- See also: CAD-REF Homepage — http://cadref.de